CLINICAL TRIAL: NCT06038019
Title: Thresholds In Food Allergy evaluaTion And predictioN, a Prospective, Multicentre Registry Study
Brief Title: Thresholds In Food Allergy evaluaTion And predictioN
Acronym: TITAN
Status: Recruiting | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: AAAAI Foundation (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: NIF-20500
Record Dates: First submitted 2023-08-18; First posted 2023-09-14 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Tree Nut Allergy; Food Allergy
Keywords: Immunotherapy; Food Allergy; Diagnosis; Prognosis
MeSH Terms: conditions — Nut Hypersensitivity; Food Hypersensitivity; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients with suspected or confirmed food allergy
  Interventions: Diagnostic Test: Oral food challenge

INTERVENTIONS:
Diagnostic Test: Oral food challenge — Patients will undergo oral food challenge with increasing amounts of food allergen

SUMMARY:
Thresholds In food allergy evaluaTion And predictioN, a prospective, observational registry. The aim is to quantify food allergy thresholds in Canada and their clinical predictors.

ELIGIBILITY:
Inclusion Criteria:

1. Suspicion or history of food allergy based on medical history, positive skin prick test, and/or serum food-specific IgE. A suggestive history is defined as typical clinical signs and/or symptoms (urticaria, angioedema, abdominal pain, vomiting, dyspnea, wheeze) within 60 minutes of the ingestion of a food.
2. Ability to discontinue all antihistamines for 1 week before oral food challenge.

Exclusion Criteria:

1. Previous desensitization treatment to a food allergen
2. Allergies to any component of the oral challenge vehicle
3. Unstable conditions including uncontrolled asthma or chronic urticaria
4. Any clinically significant disease/chronic medical condition which may interfere with study evaluations.

Ages: 3 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients suspected or confirmed to be food allergic
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2050-11-01 (Estimated); Study Completion 2051-01-01 (Estimated)

PRIMARY OUTCOMES:
Eliciting dose thresholds to food challenge | 1 year
  Threshold are measured by controlled food challenge to incremental doses of allergen (g) and are adjudicated according to CoFAR v3.0 criteria

SECONDARY OUTCOMES:
Food Allergy Quality of Life Questionnaire Child Form | 1 year
  The number of items found in the child form questionnaire includes 30 items. Food allergy quality of life questionnaire is answered on a 7-point scale (0 to 6) with higher scores representing worse impairment.
Food Allergy Quality of Life Questionnaire Teen Form | 1 year
  The number of items found in the Teen Form questionnaire includes 26 items. Food allergy quality of life questionnaire is answered on a 7-point scale (0 to 6) with higher scores representing worse impairment.
Food Allergy Quality of Life Questionnaire Adult Form | 1 year
  The number of items found in the Adult Form questionnaire includes 35 items. Food allergy quality of life questionnaire is answered on a 7-point scale (0 to 6) with higher scores representing worse impairment.
Food Allergy Quality of Life Questionnaire Parent Form | 1 year
  The number of items found in the Parent Form questionnaire includes 38 items. Food allergy quality of life questionnaire consists of 3 to 4 domains, each question is answered on a 7-point scale (0 to 6) with higher scores representing worse impairment.
Skin Prick Testing | 1 year
  Measured by mean wheal size (mm)
Specific IgE | 1 year
  Measured by ImmunoCap (kU/L)
Basophil Activation Test | 1 year
  Measured by flow cytometry (cell frequency basophils and median fluorescence intensity)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Chu, MD PhD FRCPC, Principal Investigator — Hamilton Health Sciences & McMaster University
Locations (1):
- McMaster University Medical Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Will consider on a case by case basis.